CLINICAL TRIAL: NCT06318052
Title: The Effect Of Fractional CO2 Laser Therapy On Cancer Survivors With Genitourinary Syndrome Of Menopause (GSM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUM-ABU-CO2-FemTouch-19-01
Record Dates: First submitted 2023-10-26; First posted 2024-03-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Vaginal Atrophy Patients With GSM

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CO2 laser treatment (Experimental): The FemTouch delivery system is used in conjunction with the AcuPulse CO2 laser system and the AcuScan120 microscanner to provide fractional treatments in gynecology. The system enables the delivery of laser energy along the vaginal walls. Through the use of the scanner, this laser energy is delivered in a fractional manner, selectively treating less than 100% of the tissue surface. This allows the tissue to heal much faster than when treating non-fractionally (100% of the surface) because much of the tissue is left unharmed, while the efficacy of the treatment remains significant.
  Interventions: Device: The FemTouch delivery system
- Gynomunal gel treatment (Active Comparator): Gynomunal is a hormone/free, vaginal moisturizing gel for women with vaginal dryness. Gynomunal has been clinically proven in treating vaginal dryness, and its symptoms, including itching, burning, and pain (as well as discomfort during sex). Gynomunal is a liposomal formulation containing natural hop extract, Vitamin E and hyaluronic acid.
  Interventions: Drug: Gynomunal gel treatment

INTERVENTIONS:
Device: The FemTouch delivery system — The FemTouch delivery system is used in conjunction with the AcuPulse CO2 laser system and the AcuScan120 microscanner to provide fractional treatments in gynecology
  Arms: CO2 laser treatment
Drug: Gynomunal gel treatment — hormone/free, vaginal moisturizing gel for women with vaginal dryness
  Arms: Gynomunal gel treatment

SUMMARY:
Improvement in cancer therapies has led to an increase in the number of women surviving chemotherapy (and other treatments) and overcoming cancer. This patient population presents specific clinical needs as chemotherapy (and other cancer treatments) treatment side effects can lead to early appearance of menopause symptoms and conventional hormonal treatments are contraindicated for these patients. The use of CO2 laser treatment has been shown to provide relief of Genitourinary Syndrome Of Menopause (GSM) symptoms in women and might provide a significant improvement in the quality of life for cancer survivors. The current study is designed to demonstrate the safety and efficacy of CO2 laser for treatment of GSM symptoms in cancer survivors suffering from GSM symptoms, with limited access to hormonal treatment.

DETAILED DESCRIPTION:
GSM-related symptoms significantly decrease the quality of life of post-menopausal women and harm the quality of life of up to seventy-five percent of breast cancer survivors who suffer from one or more GSM symptoms. Although varieties of hormonal and non-hormonal treatment options are available for post-menopausal women, the level of compliance is variable. One of the main reasons is the discomfort associated with the use of these measures, and in case of hormonal therapies certain risks and side effects. For cancer survivors, the possibility of having hormonal treatment must be considered against the possibility of increasing the risk of reoccurrence.

Therefore, women afflicted with GSM, whether it is age-related GSM or post-cancer GSM, are in need of additional therapeutic alternatives. Recently, supportive evidence is being gathered, showing that laser treatments to vaginal mucosa for GSM related symptoms are safe and effective. A prospective randomized comparative study comparing non-hormonal gel treatment to fractional CO2 vaginal laser treatment will contribute to optimizing treatment in this patient population

ELIGIBILITY:
Inclusion Criteria:

* Women who have had non-metastatic (M0, ≤Stage IIIA) cancer with any hormone receptor and her2 neu status who have completed cancer-related treatment>=6 months prior to enrollment with no evidence of metastasis or currently active disease
* Women currently on endocrine therapy, single agent Herceptin, or observation
* Patient-reported dyspareunia and/or vaginal dryness with the severity of >=4 on a scale from 0 (none) to 10 (most severe) that has been persistent for over >= 4 weeks and/or the inability to be sexually active due to pain
* Age 21 to 70 years
* Subjects seeking treatment of GSM
* Objective evidence of menopause: percentage of superficial vaginal epithelial cells of vaginal smear (MI) ≤ 5% and Vaginal fluid pH > 4.5 (for women within the first 3 years post-menopause)
* Normal Papanicolaou (PAP) test smear last performed as a standard of care
* Negative urine analysis
* Sexually active (having sexual intercourse at least once a month) or desire to maintain sexual activity
* Informed consent process completed and subject signed a consent form.
* Able and willing to comply with the treatment/follow-up schedule and requirements
* Patient is willing to use non-hormonal contraception method during the course of the study.

Exclusion Criteria:

* Active genital infection.
* Acute or (recurring) Urinary Tract Infection (UTI) or genital infection (e.g. Herpes or candida or (condyloma ) defined as > 2 episodes in the recent year.
* Hormonal replacement therapies (local or systemic) within the last 6 weeks.
* Pelvic Organ Prolapse (POP ≥ 2) according to the pelvic organ prolapse quantification system (may be relative).
* Prior reconstructive pelvic mesh surgery.
* Previous surgery in the treated area in the last 6 months.
* Participation in a study of another device or drug within 6 months prior to enrollment or during this study, if treatments of the vagina were involved.
* Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromise the subject safety.
* Patient is pregnant or planning to become pregnant within the next six months.

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the efficacy of fractionated CO2 laser treatments in cancer survivor patients with GSM as compared to the standard treatment | Through study completion, an average of 1 year
  Efficacy will be determined by an improvement from baseline to post-treatment in the score of the Vaginal Assessment Scale (VAS), mean of 4 items scored 0-3; 0=none 3=severe; higher score = worse condition.

SECONDARY OUTCOMES:
To demonstrate the efficacy of fractionated CO2 laser treatments in cancer survivor patients with GSM as compared to the standard treatment | Through study completion, an average of 1 year
  Efficacy of fractionated CO2 laser treatments will be determined by treatment completion rates (i.e. the number of women that complete the treatment regimen out of the randomized subjects).
To demonstrate the efficacy of fractionated CO2 laser treatments in cancer survivor patients with GSM as compared to the standard treatment. | Through study completion, an average of 1 year
  Efficacy of fractionated CO2 laser treatments will be determined by Subject Downtime evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Theden-Schow, Dr, Principal Investigator — Central study center
Locations (1):
- Frauenarztpraxis Heussweg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No